CLINICAL TRIAL: NCT04355429
Title: Efficacy of Captopril Nebulization in Covid-19 Patients Suffering of SARS CoV-2 Pneumonia. A Randomized Phase II Study
Brief Title: Efficacy of Captopril in Covid-19 Patients With Severe Acute Respiratory Syndrome (SARS) CoV-2 Pneumonia (CAPTOCOVID)
Acronym: CAPTOCOVID
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP200410
Record Dates: First submitted 2020-04-17; First posted 2020-04-21 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Pneumonia; Coronavirus Infection; COVID-19
MeSH Terms: conditions — Pneumonia; Coronavirus Infections; COVID-19 | interventions — Captopril

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAPTOPROL (Experimental): Inhalation administration by nebulization
  Interventions: Drug: captopril 25mg
- STANDARS CARE (No Intervention): According to surviving covid-Campaign guidelines

INTERVENTIONS:
Drug: captopril 25mg — Drug administration
  Other Names: Any
  Arms: CAPTOPROL

SUMMARY:
Captopril being an effective drug available in liquid preparation, administration by nebulization could be of interest for maximizing lung action and minimizing systemic side effects. Such a treatment might be used for "Covid-19" patients with pneumonia in order to avoid ARDS.

DETAILED DESCRIPTION:
Coronavirus Disease 2019 (COVID-19) is due to SARS-CoV-2 infection. The main cause of death is refractory acute respiratory distress syndrome (ARDS) secondary to SARS-CoV-2 pneumonia. The SARS-CoV-2 may have specific virulence factors to achieve mortality rates around 3%. As the SARS-CoV, virus responsible of the Severe Acute Respiratory Syndrome in 2003 (which mortality was around 10%), the SARS-CoV-2 uses angiotensin-converting enzyme 2 (ACE2) as the receptor binding domain for its spike protein making ACE2 the gateway in the alveolar epithelial cells1. Angiotensin-converting enzyme (ACE) and ACE2 are known to be present in respiratory epithelium and to have antagonist physiological functions. ACE2 has an anti-inflammatory, anti-fibrosing role, anti-oxydant and vasodilatator activity, while ACE has the opposite characteristics. These two enzymes have a negative control on each other, one inhibiting the other. Demonstrated that SARS-CoV is responsible of a downregulation of ACE2 functions by using ACE2 as cell receptor2. While ACE2 is downregulated, ACE activity increase leading to more alveolar damage and acute respiratory failure.

ACE inhibitors are common drugs used to treat hypertension worldwide. Using an ACE inhibitor as treatment against SARS-CoV-2 could be counter-intuitive because increasing ACE2 expression would open the cellular gate to the virus3,4. However, ACE2 was described as protecting lung injury2, leading Recombinant Human ACE2 as a perspective for SARS-CoV-2 treatment.

A simple way to increase ACE2 in patients with SARS-CoV-2 pneumonia could be an inhalation of ACE inhibitor.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalization for acute respiratory failure requiring oxygen administration ≥3L/mn
2. Age > 18 years or older
3. Presence of pneumonia
4. PCR SARS-CoV-2 positive in any biological sample in the last 7 days
5. Patient affiliated to social security regime
6. Written informed consent provided by the patient or alternatively by next-of-kin, or in emergency situations, prior to any protocol-specific procedures

Exclusion Criteria:

1. Decision of withholding invasive mechanical ventilation
2. Shock requiring vasopressor infusion
3. Co-infection with another respiratory pathogen which could be responsible of pneumonia
4. Hypersensitivity to captopril, to any other angiotensin converting enzyme inhibitor or any of the excipients of the specialty used
5. History of angio-oedema
6. History of ACE-inhibitor allergy
7. Known pregnancy or current lactation: Female subject of childbearing potential should have a negative serum pregnancy test prior to receiving the first dose of study medication.
8. Patient who is currently enrolled in other investigational study;
9. Persons deprived of their liberty by judicial or administrative decision,
10. Persons under legal protection/safeguard of justice,
11. Patients under duress psychiatric care,
12. Persons admitted to a health or social institution
13. Patient on state medical aid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2020-05-05 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Efficacy of captopril nebulization addition to standard of care compared to standard of care. | 14 Days
  To assess determine the efficacy of captopril nebulization addition to standard of care compared to standard of care in term of 14-day ventilation free survival

CONTACTS AND LOCATIONS:
Overall Officials: Yacine TANDJAOUI-LAMBIOTTE, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (10):
- France (10):
  - CH Victor Dupuy- Argenteuil, Argenteuil
  - Hôpital Avicenne,, Bobigny
  - Hôpital Avicenne, Bobigny
  - Hôpital Antoine Béclère, Clamart
  - CH de Compiègne-Noyon, Compiègne
  - Groupe hospitalier Sud Ile de France, Melun
  - Hôpital de la Pitié- Salpêtrière, Paris
  - Hôpital Tenon, Paris
  - CHRU de Tours, Hôpital Bretonneau, Tours
  - Hôpital de Tours, Tours

REFERENCES:
- [Background] Gurwitz D. Angiotensin receptor blockers as tentative SARS-CoV-2 therapeutics. Drug Dev Res. 2020 Aug;81(5):537-540. doi: 10.1002/ddr.21656. Epub 2020 Mar 4. PMID 32129518
- [Result] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Result] Li F, Li W, Farzan M, Harrison SC. Structure of SARS coronavirus spike receptor-binding domain complexed with receptor. Science. 2005 Sep 16;309(5742):1864-8. doi: 10.1126/science.1116480. PMID 16166518
- [Result] Imai Y, Kuba K, Rao S, Huan Y, Guo F, Guan B, Yang P, Sarao R, Wada T, Leong-Poi H, Crackower MA, Fukamizu A, Hui CC, Hein L, Uhlig S, Slutsky AS, Jiang C, Penninger JM. Angiotensin-converting enzyme 2 protects from severe acute lung failure. Nature. 2005 Jul 7;436(7047):112-6. doi: 10.1038/nature03712. PMID 16001071
- [Result] Zhang H, Penninger JM, Li Y, Zhong N, Slutsky AS. Angiotensin-converting enzyme 2 (ACE2) as a SARS-CoV-2 receptor: molecular mechanisms and potential therapeutic target. Intensive Care Med. 2020 Apr;46(4):586-590. doi: 10.1007/s00134-020-05985-9. Epub 2020 Mar 3. No abstract available. PMID 32125455